CLINICAL TRIAL: NCT00851513
Title: Therapeutic Effects Analysis of Pudendal Nerve Infiltrations After 3 Months, in Patients Suffering of Pudendal Neuralgia
Acronym: INFILTHERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRD08/6-B
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Pudendal Neuralgia; Canal Syndrome
Keywords: Pudendal neuralgia; pudendal nerve; Alcock's canal syndrome; Canal syndrome; neuropathic pain; infiltration; randomized protocol; pain scales
MeSH Terms: conditions — Pudendal Neuralgia; Neuralgia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Group B (Experimental): local anesthetics (lidocaine) associated with local steroids (depo-medrol)
  Interventions: Drug: Lidocaine; Drug: Depmedrol
- Group C (Experimental): local anesthetics (lidocaine) associated with local steroids (depomedrol) and important volumes of physiological serum
  Interventions: Drug: Lidocaine; Drug: Depmedrol; Other: physiological serum
- Group A (Active Comparator): only local anesthetic (lidocaine)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — local anesthetics
Drug: Depmedrol — local steroids
  Arms: Group B; Group C
Other: physiological serum — important volumes of physiological serum
  Arms: Group C

SUMMARY:
Pudendal neuralgia is a recent identified pathology, extremely invalidating, related to chronic pelvic entrapment. Nowadays, pudendal neuralgia can be treated with:

* neuropathic pains treatment
* specific kinesitherapy
* Alcock's canal and sacrospinal ligament infiltrations under scan
* with diagnostic block
* local steroids injections
* and surgical decompression of pudendal nerve with transrectal approach.

Only surgery was validated after a randomised protocol studying surgery versus abstention, performed and published by the CHU de Nantes. Many techniques have been proposed for realization of pudendal nerve infiltrations. The results of these infiltrations have never been published, and no randomised study had ever evaluated those results, even at short-run. Very few randomized studies have validated steroids infiltrations techniques in canal syndrome neuropathies.

The primary objective of the investigators phase IV trial is to evaluate the efficacy of three different types of pudendal nerve infiltrations in Alcock's canal and sacrospinal ligament:

* group A: only local anesthetic (control arm)
* group B: local anesthetics associated with local steroids
* group C: local anesthetics associated with local steroids and important volumes of physiological serum

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting the four indispensable clinical criteria for pudendal neuralgia (Nantes' criteria)
* Man or woman aged more than 18 years old
* Suffering from pudendal neuralgia since more than six months
* Without previous infiltration identical to the one proposed by the protocol
* Without previous surgery of pudendal nerve
* Without any hemorrhagic risk factor
* No contra-indication to Lidocaïne, Depo-medrol or contrast-product injections
* Pain intensity with an average > or = 40/100 (measured by scales during the fifteen days before infiltration)

Exclusion Criteria:

* Patient presenting one of the four exclusion clinical criterium for pudendal neuralgia (Nantes' criteria)
* Patient who has filled his "pain note book" during less than 5 days over the 15 days before the infiltration
* Pregnancy
* Depression (Beck scale > 16/39)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The main objective is to evaluate, after 3 months, the therapeutical efficacy on pain of steroids pudendal nerve infiltration, in patients suffering from pudendal neuralgia with canal syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques LABAT, Principal Investigator — Nantes University Hospital
Locations (9):
- France (9):
  - CH de la Côte Basque, Bayonne
  - Centre MARIENIA, Cambo-les-Bains
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hospices Civils de Lyon, Lyon
  - CHU de Nantes, Nantes
  - Catherine de Sienne, Nantes
  - Hôpital Rothschild, Paris
  - Scanner Saint Hilaire, Rouen
  - Hôpital Charles Nicolle, Rouen